CLINICAL TRIAL: NCT05240027
Title: To Vape or Not to Vape
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI left the site prior to providing results.
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 009.ONC.2020.D
Record Dates: First submitted 2021-11-09; First posted 2022-02-15 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Vaping
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Middle, High and College students within the Dallas-Fort Worth area that may Vape (Other): The program will be going to middle school, high school, and college campuses in the Dallas-Fort Worth (DFW) area to speak with students about vaping. The program will be implemented by community outreach, as the students will be presented with information about vaping and the resources necessary to prevent or stop vaping.
  Interventions: Behavioral: Vape use survey

INTERVENTIONS:
Behavioral: Vape use survey — pre & post test surveys

SUMMARY:
The overall goal of this study is to increase knowledge of vaping and its associated risks. This study will find the patterns of vaping, and how it all started among adolescents. Investigators want to know if students are aware of the serious and long term effects of vaping. This program titled, "To Vape or Not to Vape", will provide education to adolescents and young adults about the potential risk of vaping in an effort to assist with lowering the usage rates within the population. Content will include information about current statistics, potential short-term and long-term side-effects, and healthy alternatives for dealing with stress and peer-pressure. Investigators anticipate that this program will increase this population's knowledge about the risks of vaping products, and deter them from future use of the products. Effectiveness of this program will be measured by pre and post-tests. Investigators believe this program will make at least 50 percent of the participants more aware of the dangers and consequences of vaping, potentially lowering the rates of those participating in this habit while also preventing others from starting.

DETAILED DESCRIPTION:
The overall goal of this study is to increase knowledge of vaping and its associated risks. This study will find the patterns of vaping, and how it all started among adolescents. Investigators want to know if students are aware of the serious and long term effects of vaping. This program titled, "To Vape or Not to Vape", will provide education to adolescents and young adults about the potential risk of vaping in an effort to assist with lowering the usage rates within the population. Content will include information about current statistics, potential short-term and long-term side-effects, and healthy alternatives for dealing with stress and peer-pressure. Investigators anticipate that this program will increase this population's knowledge about the risks of vaping products, and deter them from future use of the products. Effectiveness of this program will be measured by pre and post-tests.

ELIGIBILITY:
Inclusion Criteria:

* The program's targeted population is starting at the middle school grade levels, up to college.
* Live in the DFW metroplex
* Willing to participate throughout the presentation

Exclusion Criteria:

* Less than 12 years old
* Students that are not in the DFW metroplex

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
percentage of vape users | The program will last 5 months between March 2020 and August 2020.
  Investigators will obtain the percentage of vape users and their reasons for vaping from information gathered from (per-test questionnaire).
reasons for vaping | The program will last 5 months between March 2020 and August 2020.
  Investigators will obtain the percentage of vape users and their reasons for vaping from information gathered from (per-test questionnaire).

SECONDARY OUTCOMES:
Educational Effectiveness | The program will last 5 months between March 2020 and August 2020.
  Changes in the degree of understanding will be assessed from the results of the pre and post-test (questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Maiya Bangurah, MBA, Principal Investigator — Methodist Health System Clinical Research Institute
Locations (1):
- Methodist Dallas Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-19): https://cdn.clinicaltrials.gov/large-docs/27/NCT05240027/Prot_SAP_000.pdf